CLINICAL TRIAL: NCT06429696
Title: Single-arm, Prospective Clinical Study of PD-L1 Inhibitor Combined With Apatinib as First-line Maintenance Treatment for Extensive-stage Small Cell Lung Cancer
Brief Title: PD-L1 Inhibitor Combined With Apatinib as First-line Maintenance Treatment for Extensive-stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-220
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: first-line maintenance treatment; PD-L1 inhibitor; apatinib; ES-SCLC
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 inhibitor combined with apatinib (Experimental): Six-month progression-free survival rate (6-month PFS rate) of PD-L1 inhibitor combined with apatinib in first-line maintenance treatment of extensive-stage small cell lung cancer (ES-SCLC)
  Interventions: Drug: PD-L1 inhibitor combined with apatinib

INTERVENTIONS:
Drug: PD-L1 inhibitor combined with apatinib — Every 3 weeks (21 days) is a treatment cycle. After 4-6 cycles of induction therapy, patients whose efficacy is evaluated as CR, PR or SD (according to RECIST 1.1) will enter maintenance therapy until the disease progresses and becomes intolerable. Toxic and side effects, death, withdrawal of information or the investigator's decision to withdraw the subject from the study, non-compliance with study treatment or other reasons specified in the study procedures or protocol, or treatment for up to 2 years. Maintenance treatment: PD-L1 inhibitor + apatinib 250 mg po qd, maintained for up to 2 years. Note: The specific PD-L1 inhibitor is selected by the researcher, such as adebelimab 1200mg iv, q3w; or atezolizumab 1200mg iv d1, q3w; or durvalumab 1500mg iv d1, q3w . The selection of PD-L1 inhibitors in the maintenance phase is consistent with the first-line standard treatment in the induction phase.

SUMMARY:
This is a prospective, single-arm clinical study designed to evaluate the 6-month progression-free survival rate (6-month PFS rate) of a PD-L1 inhibitor combined with apatinib as first-line maintenance treatment for extensive-stage small cell lung cancer (ES-SCLC). The study plans to recruit 40 patients. After receiving 4-6 cycles of induction therapy, patients whose efficacy is evaluated as CR, PR or SD (according to RECIST 1.1) will enter maintenance therapy with PD-L1 inhibitor + apatinib 250 mg po qd. , the selection of PD-L1 inhibitors in the maintenance phase is consistent with the first-line standard treatment in the induction phase. Efficacy was assessed using RECISIT 1.1, with imaging evaluations every 6 weeks (±7 days) for 48 weeks after the first dose and every 9 weeks (±7 days) after week 48, regardless of treatment delays or interruptions, until Disease progression or study termination, whichever occurs first. The primary efficacy endpoint of this study is 6-month PFS rate, and secondary efficacy endpoints include median PFS, median OS and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old, both men and women are welcome;
2. Extensive-stage small cell lung cancer confirmed by histology or cytology (staging according to the American Veterans Lung Cancer Association, VALG);
3. Patients whose induction therapy must receive the first-line standard treatment regimen of PD-L1 monoclonal antibody combined with chemotherapy, and whose efficacy evaluation is CR, PR or SD (according to RECIST 1.1); patients who have previously undergone surgical treatment and receive curative adjuvant therapy such as radiotherapy , chemotherapy patients, there is a treatment-free interval of at least 6 months from the last chemotherapy, radiotherapy or chemoradiotherapy to the diagnosis of extensive-stage SCLC;
4. Expected survival time ≥12 weeks;
5. ECOG physical status score 0~1 points;
6. Before the first dose of study drug, laboratory test values must meet the following conditions:

   1. Blood routine (no blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before screening): WBC ≥3.0 × 109/L; ANC ≥1.5 × 109/L; PLT ≥100 × 109/L; HGB ≥90 g/L;
   2. Liver function: AST ≤2.5 × ULN in subjects without liver metastasis; ALT ≤2.5 × ULN; ALT and AST in subjects with liver metastasis ≤5 × ULN; TBIL ≤1.5 × ULN;
   3. Renal function: serum Cr ≤1.5 × ULN or CrCl ≥50 mL/min (using Cockcroft/Gault formula);
   4. Coagulation function: INR ≤1.5 × ULN, APTT ≤1.5 × ULN (only applicable to patients who are not currently receiving anticoagulation therapy);
7. Women of childbearing age must have a serum pregnancy test within 7 days before taking the drug for the first time, and the result is negative. Female subjects of childbearing age and male subjects whose partners are women of childbearing age must agree to use contraception within 24 weeks from signing the informed consent form to the last administration of the study drug;
8. The subjects voluntarily joined this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Patients transformed from non-small cell carcinoma (NSCLC) to SCLC or SCLC with mixed histology;
2. Meningeal metastasis or symptomatic central nervous system metastasis; for patients with asymptomatic brain metastasis or stable symptoms for ≥ 2 weeks after treatment of brain metastasis, they can participate in this study as long as they meet all the following criteria: Outside the central nervous system Have measurable lesions, no metastasis to the meninges, midbrain, pons, cerebellum, medulla oblongata or spinal cord, no previous history of intracranial hemorrhage, and stop hormone therapy 14 days before the first dose of study drug;
3. Third space effusion with clinical symptoms requires repeated drainage, such as pericardial effusion, pleural effusion and peritoneal effusion that cannot be controlled by pumping or other treatments;
4. Have a history of idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, infectious pneumonia, radiation pneumonitis requiring steroid treatment, active tuberculosis, or other serious effects on the lungs Functional moderate to severe lung disease;
5. There is an active autoimmune disease and corticosteroids (>10 mg/day prednisone or equivalent dose) or other immunosuppressants are used within 14 days before the first medication;
6. Have serious cardiovascular diseases, such as New York Heart Association (NYHA) grade 2 or above heart failure, unstable angina, unstable arrhythmia, and myocardial infarction occurring within 3 months before enrollment or cerebrovascular accident;
7. Other malignant tumors ≤5 years before the first dose of medication (fully treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery can be admitted) group and allows hormone therapy for non-metastatic prostate or breast cancer);
8. Hypertension that cannot be controlled by oral antihypertensive drugs (systolic blood pressure ≧140mmHg or diastolic blood pressure ≧90mmHg);
9. Urine routine shows urine protein ≥++ and confirms that the 24-hour urine protein quantification is >1.0 g;
10. Risk of bleeding: Have clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, bleeding gastric ulcer, etc.; suffer from hereditary or acquired bleeding diseases or coagulation Functional disorders, such as aplastic anemia, etc.; taking anticoagulant or antiplatelet drugs (such as warfarin, phenprocoumon);
11. Those who have recently experienced intestinal obstruction or gastrointestinal perforation (within 3 months); or those who are unable to swallow tablets normally, which may affect drug absorption as judged by the researcher;
12. People with the following infectious diseases are not allowed to join the group:

    1. HBsAg is positive and the HBV DNA copy number is greater than the upper limit of normal value (1000 copies/ml or 500IU/ml) in the laboratory of the research center;
    2. HCV positive (HCV RNA or HCV Ab detection indicates acute or chronic infection);
    3. Known history of HIV positivity or known acquired immunodeficiency syndrome;
13. Have undergone major surgery within 28 days before the screening period, or plan to undergo major surgery during the study period;
14. Have received systemic immunosuppressive drug treatment (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide and anti-tumor necrosis factor [anti-tumor necrosis factor] within 1 week before the first medication) TNF] drugs). Patients receiving short-term, systemic immunosuppressive therapy, such as glucocorticoids for nausea, vomiting, or allergic reaction management or prophylaxis, may be enrolled in the study after approval by the investigator;
15. Live attenuated vaccines are used within 28 days before the first dose, or live attenuated vaccines are expected to be needed during the study;
16. Known to be allergic to study drugs or excipients, known to have severe allergic reactions to any monoclonal antibody drug;
17. Have received any other experimental drug treatment or participated in another interventional clinical study within 4 weeks before the first use of the drug;
18. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation;
19. According to the researcher's judgment, the subject has other factors that may lead to the forced termination of this study, such as non-compliance with the protocol, other serious diseases (including mental illness) that require combined treatment, and family or social factors that may affect the study. to the safety of subjects or the collection of information and samples

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival (PFS) | 2 years
  Defined as the time between the onset of PD when the patient first received study drug and death, whichever occurred first.

SECONDARY OUTCOMES:
Median progression-free survival (PFS) | 3 years
  Defined as the time between the onset of PD when the patient first received study drug and death, whichever occurred first.
Median overall survival (OS) | 3 years
  Defined as the time between the patient's first receipt of study drug and death
Objective response rate (ORR) | 3 years
  Defined as the proportion of patients achieving complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Wangjun Liao, MD, PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No